CLINICAL TRIAL: NCT01001624
Title: Efficacy of Melanil in the Treatment of Melasma
Brief Title: Melanil in the Treatment of Melasma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Catalysis SL (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAT-0914-CU
Record Dates: First submitted 2009-10-23; First posted 2009-10-26 (Estimated); Last update posted 2012-05-04 (Estimated); Status verified 2012-05

CONDITIONS: Melasma
Keywords: Cosmetic; Facial cream; Melasma; Melanil
MeSH Terms: conditions — Melanosis | interventions — hydroquinone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Melanil facial cream
  Interventions: Other: Melanil facial cream
- B (Active Comparator): Hydroquinone 2% cream
  Interventions: Other: Hydroquinone 2% cream

INTERVENTIONS:
Other: Melanil facial cream — Dosage commensurate with surface to be treated, Melanil facial cream (Topical use), twice a day, for 8 weeks. The affected surface will be washed and dried before application with a thin layer of Melanil facial cream.
  Arms: A
Other: Hydroquinone 2% cream — Dosage commensurate with surface to be treated, Hydroquinone 2% cream (Topical use), twice a day, for 8 weeks. The affected surface will be washed and dried before application with a thin layer of Hydroquinone 2% cream.
  Arms: B

SUMMARY:
The purpose of the study is to assess the efficacy of Melanil facial cream in the treatment of melasma. The duration of this double-blind phase 3 clinical trial will be 54 weeks. The control group will receive treatment with Hydroquinone (2%). The estimated number of subjects to be recruited and randomized for the study is 150. The primary outcome measure: Melasma Area and Severity Index (MASI) score will be assessed at the beginning of the study and at weeks 4, 8, 12 and 54. Photographs taken at the beginning of the study and at weeks 8, 12 and 54 will be evaluated by two independent dermatologists. Occurrence of adverse effects will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Melasma
* Fitzpatrick's skin types I to IV
* Signed informed consent
* Given verbal agreement on protection from UV light during treatment by the usage of physical barriers (umbrellas, caps, hats, etc).

Exclusion Criteria:

* Fitzpatrick's skin types V and VI
* Treatment with steroids within the duration of the clinical trial.
* Oral contraception within the duration of the clinical trial
* Usage of other cosmetics within the duration of the clinical trial
* Treatment with Clofazimine within the duration of the clinical trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2009-10; Primary Completion 2010-10 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
MASI score, at the beginning of the study and at weeks 4, 8 (end of the treatment), 12 and 52. | 52 weeks

SECONDARY OUTCOMES:
Occurrence of adverse effects within the 8 week treatment period and at weeks 12,24 and 52. | 52 weeks
Photographs, at the beginning of the study and at weeks 8, 12 and 52. | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo Abreu Daniel, PhD, Principal Investigator — "Cdte. Manuel Fajardo Rivero" Clinical-Surgical-Docent Hospital
Locations (1):
- "Cdte. Manuel Fajardo Rivero" Clinical-Surgical-Docent Hospital, Havana, La Habana, Cuba